CLINICAL TRIAL: NCT05632965
Title: Thyroid Function in Sick and Healthy Preterm Infants Admitted in NICU of Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Ali Nahall, Principal Investigator, Assiut University
Other Study IDs: TFPTI
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy preterm infants: Thyroid function in Preterm infants not needing hospital admission will be estimated at day 3 and day 10 of life.
- Sick preterm infants: Thyroid function in sick preterm infants admitted to NICU will be estimated at day 3 and day 10 of life .

SUMMARY:
Thyroid hormones are the cornerstones of a complex system that plays an important role in the growth and development of children, especially in the development of the nervous system and brain. Therefore, even minimal disruptions of this system can cause permanent damage.

Thyroid dysfunction is a common problem in pre-term infants. Hypothyroxinemia of prematurity within the first month of life may represent important prognostic information about morbidity and mortality. Thyroid hormone synthesis may be disrupted in co-morbid conditions . worsening the metabolism of premature infants and causing higher hormone levels compared to healthy infants.

DETAILED DESCRIPTION:
The most common thyroid function disorder in premature infants is physiological hypothyroxinemia, followed by hypothyroidism of non-thyroidal causes. In pre-maturity, several factors can inhibit the conversion of peripheral T4 to T3, including hypoxemia, acidosis, infections, hypoglycemia, hypocalcemia and malnutrition . Some rare conditions include transient secondary/tertiary hypothyroidism, transient primary hypothyroidism and permanent primary hypothyroidism.

Thyroid dysfunction has been reported to be more common in infants with low birth weight due to inadequate intrauterine nutrition, hypoxia, and acidosis.In addition, a meta-analysis found that birth weight and gestation week age closely related to thyroid function tests. Plasma T4, FT4, T3, rT3, (thyroid stimulating hormone), and (thyroxin binding globulin) concentrations during the first 8 weeks after birth in infants of 28-30 weeks gestation and in infants of <28 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants (<37w gestational age) admitted to NICU unit of assiut university children hospital with various problems as : •respiratory distress

  * hypoxia
  * sepsis
  * necrotizing enterocolitis
  * receiving TPN (total parental nutrition)
  * infants presented with jaundice.
* Another group of healthy preterm of comparable gestational age not complaining from any problems coming to routine postnatal checkup and outpatient clinic of neonatal unit will be taken .

Exclusion Criteria:

* preterm infants with : • fetal congenital malformations.

Ages: 3 Days to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: all cases of preterm infants fulfilling the inclusion criteria attending Neonatal Intensive Care unit at Assiut University children Hospital during one year.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-17 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Thyroid function | 10 days
  TSH level free T3 freeT4

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Ali, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Van Wassenaer, A., Kok, J., Dekker, F. et al. Thyroid Function in Very Preterm Infants: Influences of Gestational Age and Disease. Pediatr Res 42, 604-609 (1997). — https://doi.org/10.1203/00006450-199711000-00009